CLINICAL TRIAL: NCT05633732
Title: Echocardiography Image Quality Management System Based on Deep Learning: A Single-center Prospective Study
Brief Title: Developing Echocardiography Image Quality Management System Based on Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Southeast University, China (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-337-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-09

CONDITIONS: Echocardiography
Keywords: Echocardiography; Quality Management System; Deep learning; Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standardized View Group: The echocardiography view images of patients in this group are standardized.

SUMMARY:
To develop an echocardiography image quality management system based on deep learning to achieve objective and accurate automatic echocardiography image quality control. A total of 2000 patients performing transthoracic echocardiography were prospectively enrolled in the Department of Ultrasound Medicine of the Affiliated Drum Tower Hospital with Medical School of Nanjing University. The data of 8 TTE view segmentations were collected, including the views of the parasternal long axis of the left ventricle (PLAX_LV), parasternal short axis of the large vessel level (PSAX_GV), parasternal short axis of the mitral valve level (PSAX_MV), parasternal short axis of the papillary muscle level (PSAX_PM), parasternal short axis of the apical level (PSAX_AP), apical four cavity (A4C), apical three cavity (A3C), apical two cavity (A2C). The data of 1500 patients were used as the training set, and the rest were used as the validation set. These video data were classified into corresponding view segmentations and analyzed by the Video Swin Transformed Model. Then, the scoring module of different view segmentations combined key frame extraction, image segmentation, video target recognition and video classification model were established. At the same time, the scores achieved by the automatic echocardiography image assessment system were compared with the artificial score. By constantly correcting and learning and eventually building an primary automated grading system. At last, the automatic echocardiography image assessment system was constructed and performed on the rest 500 patients.

DETAILED DESCRIPTION:
To develop an echocardiography image quality management system based on deep learning to achieve objective and accurate automatic echocardiography image quality control. A total of 2000 patients performing transthoracic echocardiography were prospectively enrolled in the Department of Ultrasound Medicine of the Affiliated Drum Tower Hospital with Medical School of Nanjing University. The inclusion criteria: Patients with standardized TTE view segmentation; The exclusion criteria: Patients with incomplete standard segmentations. The data of 8 TTE view segmentations were collected, including the views of the parasternal long axis of the left ventricle (PLAX_LV), parasternal short axis of the large vessel level (PSAX_GV), parasternal short axis of the mitral valve level (PSAX_MV), parasternal short axis of the papillary muscle level (PSAX_PM), parasternal short axis of the apical level (PSAX_AP), apical four cavity (A4C), apical three cavity (A3C), apical two cavity (A2C). The data of 1500 patients were used as the training set, and the rest were used as the validation set. These video data were classified into corresponding view segmentations and analyzed by the Video Swin Transformed Model. Then, the scoring module of different view segmentations combined key frame extraction, image segmentation, video target recognition and video classification model were established. At the same time, the scores achieved by the automatic echocardiography image assessment system were compared with the artificial score. By constantly correcting and learning and eventually building an primary automated grading system. At last, the echocardiography image quality management system was performed on the rest 500 patients and improved.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18years, gender unlimited;
2. Patients with standardized TTE views;
3. Subjects participated in the study voluntarily and signed informed consent;

Exclusion Criteria:

1. patients wirh incomplete standard TTE views;
2. patients with poor sound transmission conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with standardized TTE views
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the score of PSAX view | 12 months
  the score of PSAX view by the echocardiography image quality management system
the score of apical view | 12 months
  the score of apical view by the echocardiography image quality management system

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thiebaut R, Thiessard F; Section Editors for the IMIA Yearbook Section on Public Health and Epidemiology Informatics. Artificial Intelligence in Public Health and Epidemiology. Yearb Med Inform. 2018 Aug;27(1):207-210. doi: 10.1055/s-0038-1667082. Epub 2018 Aug 29. PMID 30157525
- [Background] Sengupta PP, Shrestha S. Machine Learning for Data-Driven Discovery: The Rise and Relevance. JACC Cardiovasc Imaging. 2019 Apr;12(4):690-692. doi: 10.1016/j.jcmg.2018.06.030. Epub 2018 Dec 12. No abstract available. PMID 30553684
- [Background] Ueda D, Shimazaki A, Miki Y. Technical and clinical overview of deep learning in radiology. Jpn J Radiol. 2019 Jan;37(1):15-33. doi: 10.1007/s11604-018-0795-3. Epub 2018 Dec 1. PMID 30506448
- [Background] Madani A, Arnaout R, Mofrad M, Arnaout R. Fast and accurate view classification of echocardiograms using deep learning. NPJ Digit Med. 2018;1:6. doi: 10.1038/s41746-017-0013-1. Epub 2018 Mar 21. PMID 30828647